CLINICAL TRIAL: NCT03557333
Title: Open-label Study of Safety and Tolerability of Chronic Intermittent Usage for 24 or 52 Weeks of Intranasal Dihydroergotamine Mesylate (DHE) Administered Using the I123 Precision Olfactory Delivery (POD®) Device [INP104, POD-DHE] in Patients With Migraine Headache
Brief Title: Safety and Tolerability of POD-DHE (INP104) in Migraine (STOP 301)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Impel Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INP104-301
Record Dates: First submitted 2018-06-04; First posted 2018-06-15 (Actual); Results first posted 2021-02-12 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-02

CONDITIONS: Migraine Headache
MeSH Terms: conditions — Migraine Disorders | interventions — Dihydroergotamine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- INP104 (Experimental): 24-week treatment period for all participants followed by a 28-week treatment extension period for a subset of participants
  Interventions: Combination Product: INP104

INTERVENTIONS:
Combination Product: INP104 — No more than 2 doses within 24 hours, 3 doses within 7 days. 1.45 mg in a divided dose, one actuation per nostril.
  Other Names: Dihydroergotamine Mesylate (DHE) administered using the I123 Precision Olfactory Delivery (POD) Device; INP104, POD-DHE

SUMMARY:
This study consists of a 4-week screening period, a 24-week treatment period for all participants, followed by a 28-week treatment period extension (to 52 weeks in total) for a subset of at least 60 and up to 80 participants, and a 2-week post-treatment follow-up period.

DETAILED DESCRIPTION:
This is an outpatient study in people who currently suffer a minimum of 2 migraines per month. During the study, participants will be instructed to use no more than 2 doses of the study drug INP104 within a 24-hour period, or 3 doses in a 7-day period. Participants will self-administer INP104 nasally and record their migraines in an eDiary.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of migraine with or without aura, with at least 2 attacks per month for the previous 6 months.
* Participants must be in good general health, with no significant medical history (excluding migraine).
* Participants must have the ability and willingness to attend the necessary visits at the study center.
* Participants must be able to provide the written informed consent prior to entry into the study.
* Women of childbearing potential must agree to use adequate contraception (as defined in the protocol and by study personnel) during the study and for 30 days after the last dose fo the study drug.
* Male participants and their partners must agree to use effective contraception (as defined in the protocol and by study personnel) during the study and for 30 days after the last dose of the study drug. Male participants should also refrain from sperm donation for 30 days after study completion.

Exclusion Criteria:

* Subjects with trigeminal autonomic cephalalgias (including cluster headache, hemicrania syndromes and short-lasting unilateral, neuralgiform headache attacks with conjunctival injection and tearing), hemiplegic migraine, or migraine with brainstem aura (previously referred to as basilar migraines).
* Subjects with chronic migraines, medication overuse headache or other chronic headache syndromes.
* Subjects with ischemic heart disease or subjects with clinical symptoms or findings consistent with coronary artery vasospasm, including Prinzmetal's variant angina.
* Subjects with significant risk factors for coronary artery disease (CAD) including current use of nicotine-containing products, medical history of diabetes, uncontrolled hypertension (high blood pressure), known peripheral arterial disease, Raynaud's phenomenon, sepsis or vascular surgery (within 3 months prior to study start), or severely impaired hepatic or renal (kidney) function.
* Subjects with recurrent sinusitis or epistaxis.
* Subjects with a history or presence of alcoholism or drug abuse within 2 years prior to first study drug administration.
* Women who are pregnant, or planning to get pregnant, or who are lactating while participating in the study.
* Use of any medications prohibited by protocol.
* Use of >12 days per month of triptan or ergot-based medication in the 2 months prior to screening.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2018-07-13 (Actual); Primary Completion 2020-03-17 (Actual); Study Completion 2020-03-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (36):
- United States (36):
  - Synexus - Clinical Research Advantage, Inc. - Simon Williamson Clinical, PC., 832 Princeton Avenue Southwest, Birmingham, Alabama
  - Alabama Clinical Therapeutics, LLC., 52 Medical Park East Drive, Suite 203, Birmingham, Alabama
  - Synexus - Radiant Research, Inc. - Phoenix SE, 2081 West Frye Road, Chandler, Arizona
  - Synexus - Clinical Research Advantage, Inc., Central Phoenix Medical Clinic, LLC., 7600 North 15th Street, Suite 191, Phoenix, Arizona
  - Collaborative Neuroscience Network, LLC., 2600 Redondo Avenue, Suite 415, Long Beach, California
  - Excell Research, 3998 Vista Way, Oceanside, California
  - Synexus - Clinical Research Advantage, Inc. - Colorado Springs Family Practice, 2960 North Circle Drive, Suite 200, Colorado Springs, Colorado
  - Clinical Neuroscience Solutions, Inc., 5200 Belfort Road, Suite 420, Jacksonville, Florida
  - Clinical Neuroscience Solutions, Inc., 618 East South Street, Suite 100, Orlando, Florida
  - Meridien Research - Tampa, 5411 Beaumont Center Boulevard, Suite 760, Tampa, Florida
  - ENT Associates of South Florida, 4631 North Congress Avenue, Suite 200, West Palm Beach, Florida
  - Clinical Research of Central Florida, 500 East Central Avenue, Winter Haven, Florida
  - Synexus - Atlanta, 6065 Roswell Road, Suite 820, Atlanta, Georgia
  - Cedar Crosse Research Center, 800 South Wells Street, Suite M-15, Chicago, Illinois
  - Synexus - Clinical Research Advantage, Inc. - Allaw, 958C S. Kenmore Drive, Evansville, Indiana
  - Central Kentucky Research Associates, Inc., 3475 Richmond Road, 3rd Floor, Lexington, Kentucky
  - Tandem Clinical Research, LLC., 1111 Medical Center Boulevard, N513, Marrero, Louisiana
  - Synexus - Radiant Research, Inc., - Minneapolis, 7250 France Avenue South, Suite 417, Edina, Minnesota
  - StudyMetrix Research, LLC., 3862 Mexico Road, City of Saint Peters, Missouri
  - Synexus - Radiant Research, Inc. - St. Louis, 675 Old Ballas Road, Suite 103, St Louis, Missouri
  - Synexus - Clinical Research Advantage, Inc. - Omaha, 11020 Prairie Brook Road, Omaha, Nebraska
  - Synexus - Clinical Research Advantage, Inc. - Rita B. Chuang, MD, LLC., 2629 West Horizon Ridge Parkway, Suite 130, Henderson, Nevada
  - Hassman Research Institute, 175 Cross Keys Road, Suite 300B, Berlin, New Jersey
  - Integrative Clinical Trials, 3288 Ocean Avenue, Unit # MO, Brooklyn, New York
  - CNS Research Science, Inc., 80-15 164th Street, Jamaica, New York
  - Aventiv Research, 99 North Brice Road, Suite 260, Columbus, Ohio
  - OK Clinical Research, LLC., 120 North Bryant Avenue, Suite A5, Edmond, Oklahoma
  - Summit Research Network Oregon, 2701 North West Vaughn Street, Suite 350, Portland, Oregon
  - Frontier Clinical Research, LLC., 100 Ridge View Drive, Unit 4, Smithfield, Pennsylvania
  - Coastal Carolina Research Center, 9279 Medical Plaza Drive, Suite B2, North Charleston, South Carolina
  - MR - ClinSearch, LLC., 6035 Shallowford Road, Suite 109, Chattanooga, Tennessee
  - Clinical Neuroscience Solutions, Inc., 6401 Poplar Avenue, Suite 420, Memphis, Tennessee
  - FutureSearch Trials of Neurology, 5508 Parkcrest Drive, Suite 300, Austin, Texas
  - Synexus - Clinical Research Advantage, Inc. - Plano Internal Medicine Associates, PA., 6300 West Parker Road, Suite 220, Plano, Texas
  - Synexus - Radiant Research, Inc. - Salt Lake City, 5251 South Green Street, Suite 300B, Murray, Utah
  - National Clinical Research, Inc., 2809 Emerywood Parkway, Suite 140, Richmond, Virginia

REFERENCES:
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/Recalls/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 360 participants were enrolled and were dispensed INP104. Only those participants who dosed at least once with INP104 were included in the 24-Week Treatment Group, which was 354.
Groups:
- 24-Week Treatment Group: Participants in this group dosed at least once with INP104, and treated their migraine headaches as needed up to 2 times in 24 hours or up to 3 times per week with INP104, for up to 24-weeks.
Period: Overall Study
Arm/Group | 24-Week Treatment Group
Started | 354
Completed | 262
Not Completed | 92

BASELINE CHARACTERISTICS:
Arm/Group | 24-Week Treatment Group
Number analyzed (Participants) | 354
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 353
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 304
  Male | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 29
  Not Hispanic or Latino | 324
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 79
  White | 266
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 354
Mean number of migraines in 28-day baseline period [Mean (Standard Deviation); unit: number of migraines] | 4.60 (2.313)
Mean duration of migraine history [Mean (Standard Deviation); unit: years] | 19.5 (12.13)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: Number of participants with Serious Adverse Events (SAEs) whether or not related to study drug.
Time Frame: From study enrollment up to Week 26 (for the 24-Week Treatment Group) and up to Week 54 (for the 52-WeekTreatment Group)
Measure: Count of Participants; unit: Participants
Groups:
- 24-Week Treatment Group: Participants dosed with INP104 as needed for up to 24 weeks of treatment.
- 52-Week Treatment Group: This group is a subset of participants who completed 24 weeks of treatment and continued on study for up to 52 weeks of treatment.
Arm/Group | 24-Week Treatment Group | 52-Week Treatment Group
Number analyzed (Participants) | 354 | 73
Participants | 5 | 3

2. Primary Outcome: Number of Participants With Non-serious Treatment Emergent Adverse Events (AEs)
Description: Number of participants with non-serious treatment emergent adverse events (AEs), whether or not related to study drug.
Time Frame: From first use of INP104 up to Week 26 (for the 24-Week Treatment Group) and up to Week 54 (for the 52-WeekTreatment Group)
Measure: Count of Participants; unit: Participants
Arm/Group | 24-Week Treatment Group | 52-Week Treatment Group
Number analyzed (Participants) | 354 | 73
Participants | 241 | 61

3. Primary Outcome: Change in Nasal Mucosa
Description: Mean change from baseline in Quantitative Scoring Scale for Evaluation of the Nasal Mucosa (QSS-NM) score, reported at designated intervals on study. This scale was scored by otolaryngologists during routine endoscopy of the upper nasal cavity of participants. A minimum score of 0 means no issues were detected. A maximum score of 34 indicates severe issues (worse outcome).
Time Frame: Baseline up to Week 24 (for the 24-Week Treatment Group) and Baseline up to Week 52 (for the 52-WeekTreatment Group)
Population: Only those participants with assessments at baseline and at the indicated time point have data analyzed in that row.
Measure: Mean (Standard Deviation); unit: mean change in score on a scale
Arm/Group | 24-Week Treatment Group | 52-Week Treatment Group
Number analyzed (Participants) | 354 | 73
mean change in score on a scale
  Week 4: number analyzed (Participants) | 308 | 71
  Week 4 | 0.2 (1.26) | 0.0 (0.62)
  Week 8: number analyzed (Participants) | 291 | 69
  Week 8 | 0.2 (1.43) | 0.1 (0.91)
  Week 12: number analyzed (Participants) | 287 | 73
  Week 12 | 0.1 (0.93) | 0.1 (0.78)
  Week 24: number analyzed (Participants) | 261 | 70
  Week 24 | 0.1 (0.88) | 0.0 (0.79)
  Week 36: number analyzed (Participants) | 0 | 69
  Week 36 |  | -0.1 (0.68)
  Week 52: number analyzed (Participants) | 0 | 68
  Week 52 |  | -0.1 (0.61)

4. Primary Outcome: Change in Olfactory Function
Description: Mean change from baseline in olfactory function score, assessed using the University of Pennsylvania Smell Identification Test (UPSIT), and reported at designated intervals on study. The UPSIT is a 40 question scratch and sniff test of olfactory function. The minimum score of 0 indicates worst olfactory function, and the maximum score of 40 indicates the highest level of olfactory function detectable by the test.
Time Frame: Baseline up to Week 24 (for the 24-Week Treatment Group) and Baseline up to Week 52 (for the 52-WeekTreatment Group)
Population: Only those subjects with data at baseline and the indicated time point are included in the analysis for that row.
Measure: Mean (Standard Deviation); unit: mean change in score
Arm/Group | 24-Week Treatment Group | 52-Week Treatment Group
Number analyzed (Participants) | 354 | 73
mean change in score
  Week 12: number analyzed (Participants) | 280 | 72
  Week 12 | -0.48 (2.690) | -0.18 (2.573)
  Week 24: number analyzed (Participants) | 206 | 55
  Week 24 | -0.22 (2.270) | 0.03 (2.373)
  Week 36: number analyzed (Participants) | 0 | 70
  Week 36 |  | -0.13 (2.930)
  Week 52: number analyzed (Participants) | 0 | 65
  Week 52 |  | -0.80 (2.710)

ADVERSE EVENTS:
Time Frame: Week 0 to Week 24 (for the 24-Week Treatment Group) and Week 0 to Week 52 (for the 52-Week Treatment Group)
Groups:
- 24-Week Treatment Group: Participants in this group dosed at least once with INP104, and treated their migraine headaches as needed up to 2 times in 24 hours or up to 3 times per week with INP104, for up to 24 weeks.
- 52-Week Treatment Group: Participants in this group dosed at least once with INP104, and treated their migraine headaches as needed up to 2 times in 24 hours or up to 3 times per week with INP104, for up to 52 weeks. Participants in this treatment group are subset of those included in the 24-Week Treatment Group.
Arm/Group | 24-Week Treatment Group | 52-Week Treatment Group
All-Cause Mortality (participants affected / at risk) | 0/354 | 0/73
Serious Adverse Events (participants affected / at risk) | 5/354 | 3/73
Other Adverse Events (participants affected / at risk) | 241/354 | 61/73
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 24-Week Treatment Group (N=354) | 52-Week Treatment Group (N=73)
Visual impairment (Eye disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Status migrainosus (Nervous system disorders) | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 1
Ovarian mass (Reproductive system and breast disorders) | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 24-Week Treatment Group (N=354) | 52-Week Treatment Group (N=73)
Ear discomfort (Ear and labyrinth disorders) | 3 | 2
Nausea (Gastrointestinal disorders) | 28 | 8
Vomiting (Gastrointestinal disorders) | 10 | 3
Upper respiratory tract infection (Infections and infestations) | 38 | 15
Nasopharyngitis (Infections and infestations) | 30 | 10
Sinusitis (Infections and infestations) | 13 | 4
Urinary tract infection (Infections and infestations) | 9 | 5
Influenza (Infections and infestations) | 6 | 2
Pharyngitis streptococcal (Infections and infestations) | 7 | 2
Acute sinusitis (Infections and infestations) | 2 | 2
Bronchitis (Infections and infestations) | 5 | 2
Viral upper respiratory tract infection (Infections and infestations) | 7 | 2
Product package associated injury (Injury, poisoning and procedural complications) | 6 | 4
Foot fracture (Injury, poisoning and procedural complications) | 2 | 3
Procedural pain (Injury, poisoning and procedural complications) | 2 | 2
Olfactory test abnormal (Investigations) | 9 | 7 — Olfactory test abnormal events were asymptomatic decreases of 5 or more points from baseline on UPSIT score.
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 2
Dizziness (Nervous system disorders) | 8 | 4
Paraesthesia (Nervous system disorders) | 3 | 2
Somnolence (Nervous system disorders) | 2 | 2
Product taste abnormal (Product Issues) | 18 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 59 | 18
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 19 | 5
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 11 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 10 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Nasal mucosal disorder (Respiratory, thoracic and mediastinal disorders) | 6 | 2
Menopause (Social circumstances) | 2 | 2
Hypertension (Vascular disorders) | 4 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-04-26): https://cdn.clinicaltrials.gov/large-docs/33/NCT03557333/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-01): https://cdn.clinicaltrials.gov/large-docs/33/NCT03557333/SAP_001.pdf